CLINICAL TRIAL: NCT02065557
Title: A Multicenter, Randomized, Double-Blind Study of the Human Anti-TNF Monoclonal Antibody Adalimumab in Pediatric Subjects With Moderate to Severe Ulcerative Colitis
Brief Title: Efficacy and Safety of Adalimumab in Pediatric Subjects With Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M11-290; 2013-003032-77 (EudraCT Number)
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; adalimumab
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Adalimumab Induction Standard Dose (Experimental): Participants randomized to receive adalimumab 2.4 mg/kg (maximum dose of 160 mg) at Baseline and matching placebo at Week 1, 1.2 mg/kg (maximum dose of 80 mg) at Week 2, followed by 0.6 mg/kg (maximum dose of 40 mg) at Week 4 and Week 6.
  Interventions: Biological: Adalimumab; Biological: Placebo
- Adalimumab Induction High Dose (Experimental): Participants randomized to receive adalimumab 2.4 mg/kg (maximum dose of 160 mg) at Baseline and at Week 1, 1.2 mg/kg (maximum dose of 80 mg) at Week 2, followed by 0.6 mg/kg (maximum dose of 40 mg) at Week 4 and Week 6.
  Interventions: Biological: Adalimumab
- Adalimumab Induction High Dose - Open Label (Experimental): (After Amendment 4) participants assigned to open-label adalimumab 2.4 mg/kg (maximum dose of 160 mg) at Baseline and at Week 1, 1.2 mg/kg (maximum dose of 80 mg) at Week 2, followed by 0.6 mg/kg (maximum dose of 40 mg) at Week 4 and Week 6.
  Interventions: Biological: Adalimumab
- Maintenance Placebo (Placebo Comparator): (Prior to Amendment 4) participants demonstrating a clinical response per PMS (defined as a decrease in PMS ≥ 2 points and ≥ 30% from Baseline) at Week 8 randomized to maintenance placebo. Participants were to continue their blinded treatment during the maintenance period until Week 52 unless they had ≥ 2 flares and got open label rescue therapy after the second flare.
  Interventions: Biological: Adalimumab; Biological: Placebo
- Adalimumab Maintenance Standard Dose (Experimental): Participants demonstrating a clinical response per PMS (defined as a decrease in PMS ≥ 2 points and ≥ 30% from Baseline) at Week 8 randomized to adalimumab maintenance standard dose (0.6 mg/kg [maximum dose of 40 mg] every other week). Participants were to continue their blinded treatment during the maintenance period until Week 52 unless they had ≥ 2 flares and got open label rescue therapy after second flare.
  Interventions: Biological: Adalimumab
- Adalimumab Maintenance High Dose (Experimental): Participants demonstrating a clinical response per PMS (defined as a decrease in PMS ≥ 2 points and ≥ 30% from Baseline) at Week 8 randomized to adalimumab maintenance high dose (0.6 mg/kg [maximum dose of 40 mg] every week). Participants were to continue their blinded treatment during the maintenance period until Week 52 unless they had ≥ 2 flares and got open label rescue therapy after second flare.
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Subcutaneous (SC) injection
  Other Names: Humira
Biological: Placebo — Subcutaneous (SC) injection
  Arms: Adalimumab Induction Standard Dose; Maintenance Placebo

SUMMARY:
The purpose of the study is to demonstrate the efficacy and safety, and to assess the pharmacokinetics of adalimumab administered subcutaneously (SC) in pediatric subjects with moderate to severe ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UC for at least 12 weeks prior to screening, confirmed by endoscopy with biopsy.
* Active ulcerative colitis with a Mayo Score of 6 - 12 points and endoscopy subscore of 2 - 3 despite concurrent treatment with oral corticosteroids or immunosuppressants or both.

Exclusion Criteria:

* Subject with Crohn's disease (CD) or indeterminate colitis (IC).
* Current diagnosis of fulminant colitis and/or toxic megacolon.
* Subjects with disease limited to the rectum (ulcerative proctitis) during the screening endoscopy.
* Chronic recurring infections or active tuberculosis (TB).

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2014-10-13 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (60):
- United States (16):
  - Childrens Hospital LA /ID# 147452, Los Angeles, California
  - Univ California, San Francisco /ID# 120901, San Francisco, California
  - Arnold Palmer Hosp Children /ID# 120898, Orlando, Florida
  - Emory University Hospital /ID# 121858, Atlanta, Georgia
  - Children's Ctr Digestive, US /ID# 121855, Atlanta, Georgia
  - University of Chicago /ID# 120904, Chicago, Illinois
  - Loyola University Medical Ctr /ID# 120900, Maywood, Illinois
  - Indiana University /ID# 120908, Indianapolis, Indiana
  - Massachusetts General Hospital /ID# 124551, Boston, Massachusetts
  - Boston Childrens Hospital /ID# 147714, Boston, Massachusetts
  - Mayo Clinic - Rochester /ID# 121056, Rochester, Minnesota
  - Minnesota Gastroenterology P.A /ID# 120895, Saint Paul, Minnesota
  - Goryeb Chidlren's Hospital /ID# 121860, Morristown, New Jersey
  - North Shore University Hospital /ID# 120905, New Hyde Park, New York
  - Univ Rochester Med Ctr /ID# 127776, Rochester, New York
  - Multicare Institute for Research and Innovation /ID# 147716, Tacoma, Washington
- Womens and Childrens Hospital /ID# 127538, Adelaide, South Australia, Australia
- Austria (2):
  - Medizinische Universitat Wien /ID# 120802, Vienna, Vienna
  - LKH Salzburg and Paracelsus /ID# 123457, Salzburg
- Belgium (3):
  - UZ Brussel /ID# 120798, Jette, Brussels Capital
  - Cliniques Universitaires Saint Luc /ID# 120797, Woluwe-Saint-Lambert, Brussels Capital
  - Hosp Univ Enfants Reine Fabiol /ID# 120795, Brussels
- London Health Sciences Centre /ID# 127777, London, Ontario, Canada
- Czechia (2):
  - Palacky University /ID# 131388, Olomouc
  - Univ Hosp, Plzen, CZ /ID# 120813, Pilsen
- Hungary (2):
  - Petz Aladar Megyei Oktato Korh /ID# 124323, Győr
  - Balassa Janos County Hospital /ID# 128474, Szekszárd
- Israel (7):
  - Soroka Medical Ctr /ID# 147338, Beersheba
  - Assaf Harofeh Medical Center /ID# 147791, Be’er Ya‘aqov
  - Rambam Health Care Campus /ID# 120827, Haifa
  - Shaare Zedek Medical Center /ID# 120830, Jerusalem
  - Schneider Childrens Med Ctr /ID# 120821, Petah Tikva
  - Sheba Medical Center /ID# 124324, Ramat Gan
  - Kaplan Medical Center /ID# 150245, Rehovot
- Japan (11):
  - Kurume University Hospital /ID# 125476, Kurume-shi, Fukuoka
  - Gunma University Hospital /ID# 126345, Maebashi, Gunma
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 124482, Sapporo, Hokkaido
  - The Hospital of Hyogo College of Medicine /ID# 131665, Nishinomiya-shi, Hyōgo
  - Saiseikai Yokohamashi Tobu /ID# 124486, Yokohama, Kanagawa
  - Yokohama City Univ Medical Ctr /ID# 147763, Yokohama, Kanagawa
  - Miyagi Children's Hospital /ID# 125475, Sendai, Miyagi
  - Saitama Children's Medical Center /ID# 124485, Saitama-shi, Saitama
  - Juntendo University Hospital /ID# 124536, Bunkyo-ku, Tokyo
  - National Center for Child Health and Development /ID# 125203, Setagaya-ku, Tokyo
  - Osaka General Medical Center /ID# 124535, Osaka
- Canterbury District Health Boa /ID# 120837, Christchurch, New Zealand
- Poland (5):
  - Uni Szpital Dzieciecy w Krakowie /ID# 120915, Krakow, Lesser Poland Voivodeship
  - Centrum Zdrowia MDM /ID# 120910, Warsaw, Masovian Voivodeship
  - Gabinet Lekarski Bartosz Korcz /ID# 120916, Rzeszów
  - Samodzielny Publiczny Szpital /ID# 120839, Wroclaw
  - Polish Mothers Memorial Hosp /ID# 148497, Lodz, Łódź Voivodeship
- Slovakia (3):
  - FN s poliklinikou F.D. Rooseve /ID# 120847, Banská Bystrica
  - Univerzitna Nemocnica Bratislava /ID# 120842, Bratislava
  - Univerzitna nemocnica Martin /ID# 120844, Martin, Žilina Region
- Spain (2):
  - Hospital Univ Vall d'Hebron /ID# 120856, Barcelona
  - Hospital Infantil Universitario Nino Jesus /ID# 121862, Madrid
- United Kingdom (4):
  - The Royal London Hospital /ID# 120861, London, London, City of
  - The Royal Free Hospital /ID# 123142, London, London, City of
  - Royal Hosp for Sick Children /ID# 120864, Glasgow
  - Manchester Royal Infirmary, Ma /ID# 120862, Manchester

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Croft NM, Faubion WA Jr, Kugathasan S, Kierkus J, Ruemmele FM, Shimizu T, Mostafa NM, Venetucci M, Finney-Hayward T, Sanchez Gonzalez Y, Bereswill M, Lazar A, Turner D. Efficacy and safety of adalimumab in paediatric patients with moderate-to-severe ulcerative colitis (ENVISION I): a randomised, controlled, phase 3 study. Lancet Gastroenterol Hepatol. 2021 Aug;6(8):616-627. doi: 10.1016/S2468-1253(21)00142-4. Epub 2021 Jun 19. PMID 34153231
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prior to Protocol Amendment 4, participants were randomized 3:2 at baseline to adalimumab induction high dose or adalimumab induction standard dose. At Week 8, those demonstrating a clinical response per Partial Mayo Score (PMS) were randomized 2:2:1 to adalimumab maintenance standard dose, adalimumab maintenance high dose, or maintenance placebo.
Pre-assignment Details: After Protocol Amendment 4, participants received adalimumab induction high dose open-label. At Week 8, those demonstrating a clinical response per PMS were randomized in a 1:1 ratio to adalimumab maintenance standard dose or adalimumab maintenance high dose. "Integrated Study" data includes data from both the Main Study and the Japan Sub-Study.
Groups:
- Integrated Study: Induction Standard Dose (I-SD): Participants randomized to receive adalimumab 2.4 mg/kg (maximum dose of 160 mg) at Baseline and matching placebo at Week 1, 1.2 mg/kg (maximum dose of 80 mg) at Week 2, followed by 0.6 mg/kg (maximum dose of 40 mg) at Week 4 and Week 6.
- Integrated Study: Induction High Dose (I-HD): Participants randomized to receive adalimumab 2.4 mg/kg (maximum dose of 160 mg) at Baseline and at Week 1, 1.2 mg/kg (maximum dose of 80 mg) at Week 2, followed by 0.6 mg/kg (maximum dose of 40 mg) at Week 4 and Week 6.
- Integrated Study: Induction High Dose Open Label (I-HD-OL): (After Amendment 4) participants assigned to open-label adalimumab 2.4 mg/kg (maximum dose of 160 mg) at Baseline and at Week 1, 1.2 mg/kg (maximum dose of 80 mg) at Week 2, followed by 0.6 mg/kg (maximum dose of 40 mg) at Week 4 and Week 6.
- Integrated Study: Maintenance Placebo (M-PL): (Prior to Amendment 4) participants demonstrating a clinical response per PMS (defined as a decrease in PMS ≥ 2 points and ≥ 30% from Baseline) at Week 8 randomized to maintenance placebo. Participants were to continue their blinded treatment during the maintenance period until Week 52 unless they had ≥ 2 flares and got open label rescue therapy after the second flare.
- Integrated Study: Maintenance Standard Dose (M-SD): Participants demonstrating a clinical response per PMS (defined as a decrease in PMS ≥ 2 points and ≥ 30% from Baseline) at Week 8 randomized to adalimumab maintenance standard dose (0.6 mg/kg [maximum dose of 40 mg] every other week [eow]). Participants were to continue their blinded treatment during the maintenance period until Week 52 unless they had ≥ 2 flares and got open label rescue therapy after the second flare.
- Integrated Study: Maintenance High Dose (M-HD): Participants demonstrating a clinical response per PMS (defined as a decrease in PMS ≥ 2 points and ≥ 30% from Baseline) at Week 8 randomized to adalimumab maintenance high dose (0.6 mg/kg [maximum dose of 40 mg] every week [ew]). Participants were to continue their blinded treatment during the maintenance period until Week 52 unless they had ≥ 2 flares and got open label rescue therapy after the second flare.
Period: Induction Period
Arm/Group | Integrated Study: Induction Standard Dose (I-SD) | Integrated Study: Induction High Dose (I-HD) | Integrated Study: Induction High Dose Open Label (I-HD-OL) | Integrated Study: Maintenance Placebo (M-PL) | Integrated Study: Maintenance Standard Dose (M-SD) | Integrated Study: Maintenance High Dose (M-HD)
Started | 32 | 51 | 18 | 0 | 0 | 0
Enrolled in Main Study | 30 | 47 | 16 | 0 | 0 | 0
Enrolled in Japan Sub-study | 2 | 4 | 2 | 0 | 0 | 0
Completed | 22 | 43 | 16 | 0 | 0 | 0
Not Completed | 10 | 8 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Requires Alternative/Prohibited Therapy | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Non-Responder at Week 8 | 4 | 4 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0
Period: Maintenance Period
Arm/Group | Integrated Study: Induction Standard Dose (I-SD) | Integrated Study: Induction High Dose (I-HD) | Integrated Study: Induction High Dose Open Label (I-HD-OL) | Integrated Study: Maintenance Placebo (M-PL) | Integrated Study: Maintenance Standard Dose (M-SD) | Integrated Study: Maintenance High Dose (M-HD)
Started | 0 | 0 | 0 | 12 | 33 | 36
Completed (Completed Week 52) | 0 | 0 | 0 | 11 | 25 | 32
Not Completed | 0 | 0 | 0 | 1 | 8 | 4
Not completed — Requires Alternative/Prohibited Therapy | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 5 | 2
Not completed — Subject Non-Compliance | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Integrated Study (Main + Japan Sub- Study): I-SD: Participants randomized to receive adalimumab 2.4 mg/kg (maximum dose of 160 mg) at Baseline and matching placebo at Week 1, 1.2 mg/kg (maximum dose of 80 mg) at Week 2, followed by 0.6 mg/kg (maximum dose of 40 mg) at Week 4 and Week 6.
- Integrated Study (Main + Japan Sub- Study): I-HD: Participants randomized to receive adalimumab 2.4 mg/kg (maximum dose of 160 mg) at Baseline and at Week 1, 1.2 mg/kg (maximum dose of 80 mg) at Week 2, followed by 0.6 mg/kg (maximum dose of 40 mg) at Week 4 and Week 6.
- Integrated Study (Main + Japan Sub- Study): I-HD-OL: (After Amendment 4) participants assigned to open-label adalimumab 2.4 mg/kg (maximum dose of 160 mg) at Baseline and at Week 1, 1.2 mg/kg (maximum dose of 80 mg) at Week 2, followed by 0.6 mg/kg (maximum dose of 40 mg) at Week 4 and Week 6.
- Total: Total of all reporting groups
Arm/Group | Integrated Study (Main + Japan Sub- Study): I-SD | Integrated Study (Main + Japan Sub- Study): I-HD | Integrated Study (Main + Japan Sub- Study): I-HD-OL | Total
Number analyzed (Participants) | 32 | 51 | 18 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (2.66) | 13.8 (3.06) | 13.8 (2.82) | 14.1 (2.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 23 | 13 | 51
  Male | 17 | 28 | 5 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 28 | 45 | 15 | 88
  Black | 1 | 2 | 0 | 3
  Asian | 3 | 4 | 2 | 9
  Multiple | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4
  Japanese | 2 | 4 | 2 | 8
  No Ethnicity | 29 | 45 | 15 | 89
Full Mayo Score (FMS) [Mean (Standard Deviation); unit: score on a scale] — The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy, and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease).
  score on a scale | 7.8 (1.22) | 7.7 (1.25) | 7.7 (1.09) | 7.8 (1.20)
Partial Mayo Score (PMS) [Mean (Standard Deviation); unit: score on a scale] — The PMS (Mayo score without endoscopy) ranges from 0 (normal or inactive disease) to 9 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease).
  score on a scale | 5.7 (1.14) | 5.5 (1.24) | 5.5 (1.06) | 5.6 (1.17)
Endoscopy Subscore [Mean (Standard Deviation); unit: score on a scale] — The endoscopy subscore of the FMS ranges from 0 (normal) to 3 (severe disease).
  score on a scale | 2.1 (0.34) | 2.2 (0.40) | 2.2 (0.43) | 2.2 (0.38)
Rectal Bleeding Subscore [Mean (Standard Deviation); unit: score on a scale] — The rectal bleeding subscore of the FMS ranges from 0 (normal) to 3 (severe disease).
  score on a scale | 1.4 (0.93) | 1.5 (0.88) | 1.4 (0.97) | 1.5 (0.91)
Physicians Global Assessment Subscore [Mean (Standard Deviation); unit: score on a scale] — The physicians global assessment subscore of the FMS ranges from 0 (normal) to 3 (severe disease).
  score on a scale | 2.2 (0.40) | 2.2 (0.43) | 2.2 (0.38) | 2.2 (0.41)
Stool Frequency Subscore [Mean (Standard Deviation); unit: score on a scale] — The stool frequency subscore of the FMS ranges from 0 (normal) to 3 (severe disease).
  score on a scale | 2.1 (0.78) | 1.8 (0.88) | 1.9 (0.73) | 1.9 (0.83)

OUTCOME MEASURES:

1. Primary Outcome: Co-Primary Endpoint 1: Percentage of Participants Who Achieved Clinical Remission as Measured by Partial Mayo Score (PMS) at Week 8 - Induction Period
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The PMS (Mayo score without endoscopy) ranges from 0 (normal or inactive disease) to 9 (severe disease) and is calculated as the sum of 3 sub scores (stool frequency, rectal bleeding and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in PMS indicates improvement. Clinical remission was defined as a PMS ≤ 2 and no individual subscore > 1.
Time Frame: Week 8
Population: Intent-to-Treat (ITT): all participants who received at least 1 dose of study drug during the Induction period; analyzed as enrolled/randomized. Non-responder imputation (NRI): missing data is imputed as not having met the endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Main Study: I-SD; Integrated Study (Main + Japan Sub-Study): I-SD: Participants randomized to receive adalimumab 2.4 mg/kg (maximum dose of 160 mg) at Baseline and matching placebo at Week 1, 1.2 mg/kg (maximum dose of 80 mg) at Week 2, followed by 0.6 mg/kg (maximum dose of 40 mg) at Week 4 and Week 6.
- Main Study: I-HD; Integrated Study (Main + Japan Sub-Study): I-HD: Participants randomized to receive adalimumab 2.4 mg/kg (maximum dose of 160 mg) at Baseline and at Week 1, 1.2 mg/kg (maximum dose of 80 mg) at Week 2, followed by 0.6 mg/kg (maximum dose of 40 mg) at Week 4 and Week 6.
- Main Study: I-SD + I-HD; Integrated Study (Main + Japan Sub-Study): I-SD + I-HD: Combined I-SD + I-HD arms (see above).
- Main Study: I-HD-OL; Integrated Study (Main + Japan Sub-Study): I-HD-OL: (After Amendment 4) participants assigned to open-label adalimumab 2.4 mg/kg (maximum dose of 160 mg) at Baseline and at Week 1, 1.2 mg/kg (maximum dose of 80 mg) at Week 2, followed by 0.6 mg/kg (maximum dose of 40 mg) at Week 4 and Week 6.
Arm/Group | Main Study: I-SD | Main Study: I-HD | Main Study: I-SD + I-HD | Main Study: I-HD-OL | Integrated Study (Main + Japan Sub-Study): I-SD | Integrated Study (Main + Japan Sub-Study): I-HD | Integrated Study (Main + Japan Sub-Study): I-SD + I-HD | Integrated Study (Main + Japan Sub-Study): I-HD-OL
Number analyzed (Participants) | 30 | 47 | 77 | 16 | 32 | 51 | 83 | 18
percentage of participants | 43.3 [25.46 to 62.57] | 59.6 [44.27 to 73.63] | 53.2 [41.52 to 64.71] | 68.8 [41.34 to 88.98] | 40.6 [23.70 to 59.36] | 58.8 [44.17 to 72.42] | 51.8 [40.56 to 62.92] | 66.7 [40.99 to 86.66]
Statistical Analysis 1: Comparison: Main Study: I-SD + I-HD; Efficacy analysis was based on the Intent-To-Treat-Efficacy (ITT-E) population for the induction period. The ITT-E population was a subpopulation of the ITT population, which consisted of all participants who received at least one SC injection of the study medication during the induction period. Participants who received open-label high induction dose, because they enrolled after Protocol Amendment 4 was released, were excluded from the ITT-E population; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, rejective multiple test procedure — Adjusted p-value from a sequentially rejective multiple test procedure, testing co-primary and ranked secondary endpoints 1st for I-SD+I-HD, then for individual adalimumab dose groups (I-HD, I-SD) against the respective external placebo rate (19.83%); controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 2: Comparison: Main Study: I-HD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, rejective multiple test procedure — [p-value comment as in outcome 1, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 3: Comparison: Main Study: I-SD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p = 0.382, rejective multiple test procedure — [p-value comment as in outcome 1, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 4: Comparison: Integrated Study (Main + Japan Sub-Study): I-SD + I-HD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, rejective multiple test procedure — [p-value comment as in outcome 1, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 5: Comparison: Integrated Study (Main + Japan Sub-Study): I-HD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, rejective multiple test procedure — [p-value comment as in outcome 1, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 6: Comparison: Integrated Study (Main + Japan Sub-Study): I-SD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p = 0.344, rejective multiple test procedure — [p-value comment as in outcome 1, analysis 1]; controlling familywise Type I error of 5% in a strong sense

2. Primary Outcome: Co-Primary Endpoint 2: Percentage of Participants With Clinical Remission Per Full Mayo Score (FMS) at Week 52 in Week 8 Responders Per PMS - Maintenance Period
Description: The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy, and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). The PMS (Mayo score without endoscopy) ranges from 0 (normal or inactive disease) to 9 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding and physician's global assessment). Negative changes indicate improvement. PMS responders are defined as those with a decrease in PMS ≥ 2 points and ≥ 30% from Baseline. Clinical remission per FMS is defined as Mayo Score ≤ 2 and no individual subscore > 1.
Time Frame: Week 52
Population: Modified intent-to-treat (mITT): all Week 8 PMS responders who were re-randomized at Week 8 and received at least 1 dose of study drug during the Maintenance period; analyzed as randomized at the beginning of the Maintenance phase. NRI: missing data is imputed as not having met the endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Main Study: M-PL; Integrated Study (Main + Japan Sub-Study): M-PL: (Prior to Amendment 4) participants demonstrating a clinical response per PMS (defined as a decrease in PMS ≥ 2 points and ≥ 30% from Baseline) at Week 8 randomized to maintenance placebo. Participants were to continue their blinded treatment during the maintenance period until Week 52 unless they had ≥ 2 flares and got open label adalimumab rescue therapy after the second flare.
- Main Study: M-SD; Integrated Study (Main + Japan Sub-Study): M-SD: Participants demonstrating a clinical response per PMS (defined as a decrease in PMS ≥ 2 points and ≥ 30% from Baseline) at Week 8 randomized to adalimumab maintenance standard dose (0.6 mg/kg [maximum dose of 40 mg] eow). Participants were to continue their blinded treatment during the maintenance period until Week 52 unless they had ≥ 2 flares and got open label rescue therapy after the second flare.
- Main Study: M-HD; Integrated Study (Main + Japan Sub-Study): M-HD: Participants demonstrating a clinical response per PMS (defined as a decrease in PMS ≥ 2 points and ≥ 30% from Baseline) at Week 8 randomized to adalimumab maintenance high dose (0.6 mg/kg [maximum dose of 40 mg] ew). Participants were to continue their blinded treatment during the maintenance period until Week 52 unless they had ≥ 2 flares and got open label rescue therapy after the second flare.
- Main Study: M-SD + M-HD; Integrated Study (Main + Japan Sub-Study): M-SD + M-HD: Combined M-SD + M-HD arms (see above).
Arm/Group | Main Study: M-PL | Main Study: M-SD | Main Study: M-HD | Main Study: M-SD + M-HD | Integrated Study (Main + Japan Sub-Study): M-PL | Integrated Study (Main + Japan Sub-Study): M-SD | Integrated Study (Main + Japan Sub-Study): M-HD | Integrated Study (Main + Japan Sub-Study): M-SD + M-HD
Number analyzed (Participants) | 12 | 31 | 31 | 62 | 12 | 33 | 35 | 68
percentage of participants | 33.3 [9.92 to 65.11] | 29.0 [14.22 to 48.04] | 45.2 [27.32 to 63.97] | 37.1 [25.16 to 50.31] | 33.3 [9.92 to 65.11] | 27.3 [13.30 to 45.52] | 42.9 [26.32 to 60.65] | 35.3 [24.08 to 47.83]
Statistical Analysis 1: Comparison: Main Study: M-SD + M-HD; Efficacy analysis was based on the modified Intent-To-Treat-Efficacy (mITT-E) population for the maintenance period. The mITT-E population was a subpopulation of the mITT population, where participants in M-PL arm were excluded; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, rejective multiple test procedure — Adjusted p-value from a sequentially rejective multiple test procedure, testing co-primary and ranked secondary endpoints 1st for M-SD+M-HD, then for individual adalimumab dose groups (M-HD, M-SD) against the respective external placebo rate (18.37%); controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 2: Comparison: Main Study: M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, rejective multiple test procedure — [p-value comment as in outcome 2, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 3: Comparison: Main Study: M-SD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p = 0.382, rejective multiple test procedure — [p-value comment as in outcome 2, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 4: Comparison: Integrated Study (Main + Japan Sub-Study): M-SD + M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, rejective multiple test procedure — [p-value comment as in outcome 2, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 5: Comparison: Integrated Study (Main + Japan Sub-Study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, rejective multiple test procedure — [p-value comment as in outcome 2, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 6: Comparison: Integrated Study (Main + Japan Sub-Study): M-SD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p = 0.344, rejective multiple test procedure — [p-value comment as in outcome 2, analysis 1]; controlling familywise Type I error of 5% in a strong sense

3. Secondary Outcome: Ranked Secondary Endpoint 1: Percentage of Participants With Clinical Response Per FMS at Week 52 in Week 8 Responders Per PMS - Maintenance Period
Description: The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy, and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). The PMS (Mayo score without endoscopy) ranges from 0 (normal or inactive disease) to 9 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding and physician's global assessment). Negative changes indicate improvement. PMS responders are defined as those with a decrease in PMS ≥ 2 points and ≥ 30% from Baseline. Clinical response per FMS is defined as a decrease in FMS ≥ 3 points and ≥ 30% from Baseline.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main Study: M-PL | Main Study: M-SD | Main Study: M-HD | Main Study: M-SD + M-HD | Integrated Study (Main + Japan Sub-Study): M-PL | Integrated Study (Main + Japan Sub-Study): M-SD | Integrated Study (Main + Japan Sub-Study): M-HD | Integrated Study (Main + Japan Sub-Study): M-SD + M-HD
Number analyzed (Participants) | 12 | 31 | 31 | 62 | 12 | 33 | 35 | 68
percentage of participants | 33.3 [9.92 to 65.11] | 61.3 [42.19 to 78.15] | 67.7 [48.63 to 83.32] | 64.5 [51.34 to 76.26] | 33.3 [9.92 to 65.11] | 57.6 [39.22 to 74.52] | 65.7 [47.79 to 80.87] | 61.8 [49.18 to 73.29]
Statistical Analysis 1: Comparison: Main Study: M-SD + M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, rejective multiple test procedure — Adjusted p-value from a sequentially rejective multiple test procedure, testing co-primary and ranked secondary endpoints 1st for M-SD+M-HD, then for individual adalimumab dose groups (M-HD, M-SD) against the respective external placebo rate (26.10%); controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 2: Comparison: Main Study: M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, Chi-squared — [p-value comment as in outcome 3, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 3: Comparison: Main Study: M-SD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p = 0.008, Chi-squared — [p-value comment as in outcome 3, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 4: Comparison: Integrated Study (Main + Japan Sub-Study): M-SD + M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, rejective multiple test procedure — [p-value comment as in outcome 3, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 5: Comparison: Integrated Study (Main + Japan Sub-Study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, rejective multiple test procedure — [p-value comment as in outcome 3, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 6: Comparison: Integrated Study (Main + Japan Sub-Study): M-SD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p = 0.038, rejective multiple test procedure — [p-value comment as in outcome 3, analysis 1]; controlling familywise Type I error of 5% in a strong sense

4. Secondary Outcome: Ranked Secondary Endpoint 2: Percentage of Participants With Mucosal Healing at Week 52 in Week 8 Responders Per PMS - Maintenance Period
Description: The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy, and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). The PMS (Mayo score without endoscopy) ranges from 0 (normal or inactive disease) to 9 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding and physician's global assessment). Negative changes indicate improvement. PMS responders are defined as those participants with a decrease in PMS ≥ 2 points and ≥ 30% from Baseline. Mucosal healing per Mayo endoscopy subscore is defined as a subscore of ≤ 1.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main Study: M-PL | Main Study: M-SD | Main Study: M-HD | Main Study: M-SD + M-HD | Integrated Study (Main + Japan Sub-Study): M-PL | Integrated Study (Main + Japan Sub-Study): M-SD | Integrated Study (Main + Japan Sub-Study): M-HD | Integrated Study (Main + Japan Sub-Study): M-SD + M-HD
Number analyzed (Participants) | 12 | 31 | 31 | 62 | 12 | 33 | 35 | 68
percentage of participants | 33.3 [9.92 to 65.11] | 38.7 [21.85 to 57.81] | 51.6 [33.06 to 69.85] | 45.2 [32.48 to 58.32] | 33.3 [9.92 to 65.11] | 36.4 [20.40 to 54.88] | 48.6 [31.38 to 66.01] | 42.6 [30.72 to 55.23]
Statistical Analysis 1: Comparison: Main Study: M-SD + M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, rejective multiple test procedure — Adjusted p-value from a sequentially rejective multiple test procedure, testing co-primary and ranked secondary endpoints 1st for M-SD+M-HD, then for individual adalimumab dose groups (M-HD, M-SD) against the respective external placebo rate (22.03%); controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 2: Comparison: Main Study: M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, rejective multiple test procedure — [p-value comment as in outcome 4, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 3: Comparison: Main Study: M-SD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p = 0.382, rejective multiple test procedure — [p-value comment as in outcome 4, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 4: Comparison: Integrated Study (Main + Japan Sub-Study): M-SD + M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, rejective multiple test procedure — [p-value comment as in outcome 4, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 5: Comparison: Integrated Study (Main + Japan Sub-Study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, rejective multiple test procedure — [p-value comment as in outcome 4, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 6: Comparison: Integrated Study (Main + Japan Sub-Study): M-SD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p = 0.344, rejective multiple test procedure — [p-value comment as in outcome 4, analysis 1]; controlling familywise Type I error of 5% in a strong sense

5. Secondary Outcome: Ranked Secondary Endpoint 3: Percentage of Participants With Clinical Remission Per FMS at Week 52 in Week 8 Remitters Per PMS - Maintenance Period
Description: The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy, and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). The PMS (Mayo score without endoscopy) ranges from 0 (normal or inactive disease) to 9 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding and physician's global assessment). Negative changes indicate improvement. PMS remitters are defined as those participants with a PMS ≤ 2 and no individual subscore > 1. Clinical remission per FMS is defined as Mayo Score ≤ 2 and no individual subscore > 1.
Time Frame: Week 52
Population: Modified intent-to-treat (mITT): all Week 8 PMS responders who were re-randomized at Week 8 and received at least 1 dose of study drug during the Maintenance period; analyzed as randomized at the beginning of the Maintenance phase. Participants who were also Week 8 remitters. NRI: missing data is imputed as not having met the endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main Study: M-PL | Main Study: M-SD | Main Study: M-HD | Main Study: M-SD + M-HD | Integrated Study (Main + Japan Sub-Study): M-PL | Integrated Study (Main + Japan Sub-Study): M-SD | Integrated Study (Main + Japan Sub-Study): M-HD | Integrated Study (Main + Japan Sub-Study): M-SD + M-HD
Number analyzed (Participants) | 8 | 21 | 22 | 43 | 8 | 21 | 25 | 46
percentage of participants | 37.5 [8.52 to 75.51] | 42.9 [21.82 to 65.98] | 45.5 [24.39 to 67.79] | 44.2 [29.08 to 60.12] | 37.5 [8.52 to 75.51] | 42.9 [21.82 to 65.98] | 44.0 [24.40 to 65.07] | 43.5 [28.93 to 58.89]
Statistical Analysis 1: Comparison: Main Study: M-SD + M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, rejective multiple test procedure — Adjusted p-value from a sequentially rejective multiple test procedure, testing co-primary and ranked secondary endpoints 1st for M-SD+M-HD, then for individual adalimumab dose groups (M-HD, M-SD) against the respective external placebo rate (14.79%); controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 2: Comparison: Main Study: M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, rejective multiple test procedure — [p-value comment as in outcome 5, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 3: Comparison: Main Study: M-SD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p = 0.292, rejective multiple test procedure — [p-value comment as in outcome 5, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 4: Comparison: Integrated Study (Main + Japan Sub-Study): M-SD + M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, rejective multiple test procedure — [p-value comment as in outcome 5, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 5: Comparison: Integrated Study (Main + Japan Sub-Study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p < 0.001, rejective multiple test procedure — [p-value comment as in outcome 5, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 6: Comparison: Integrated Study (Main + Japan Sub-Study): M-SD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p = 0.292, rejective multiple test procedure — [p-value comment as in outcome 5, analysis 1]; controlling familywise Type I error of 5% in a strong sense

6. Secondary Outcome: Ranked Secondary Endpoint 4: Percentage of Participants With Corticosteroid-Free Clinical Remission Per FMS at Week 52 in Week 8 Responders Per PMS - Maintenance Period
Description: The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy, and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). The PMS (Mayo score without endoscopy) ranges from 0 (normal or inactive disease) to 9 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding and physician's global assessment). Negative changes indicate improvement. PMS responders are defined as those with a decrease in PMS ≥ 2 points and ≥ 30% from baseline. Among participants receiving systemic corticosteroids at Baseline, corticosteroid-free clinical remission per FMS at Week 52 is defined as having discontinued systemic corticosteroids prior to Week 52 and being in FMS clinical remission at Week 52 (defined as Mayo Score ≤ 2 and no individual subscore > 1).
Time Frame: Week 52
Population: mITT: all Week 8 PMS responders who were re-randomized at Week 8 and received at least 1 dose of study drug during the Maintenance period; analyzed as randomized at the beginning of the Maintenance phase. Participants receiving systemic corticosteroids at baseline. NRI: missing data is imputed as not having met the endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main Study: M-PL | Main Study: M-SD | Main Study: M-HD | Main Study: M-SD + M-HD | Integrated Study (Main + Japan Sub-Study): M-PL | Integrated Study (Main + Japan Sub-Study): M-SD | Integrated Study (Main + Japan Sub-Study): M-HD | Integrated Study (Main + Japan Sub-Study): M-SD + M-HD
Number analyzed (Participants) | 5 | 13 | 16 | 29 | 5 | 15 | 17 | 32
percentage of participants | 40.0 [5.27 to 85.34] | 30.8 [9.09 to 61.43] | 31.3 [11.02 to 58.66] | 31.0 [15.28 to 50.83] | 40.0 [5.27 to 85.34] | 26.7 [7.79 to 55.10] | 35.3 [14.21 to 61.67] | 31.3 [16.12 to 50.01]
Statistical Analysis 1: Comparison: Main Study: M-SD + M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p = 0.382, rejective multiple test procedure — Adjusted p-value from a sequentially rejective multiple test procedure, testing co-primary and ranked secondary endpoints 1st for M-SD+M-HD, then for individual adalimumab dose groups (M-HD, M-SD) against the respective external placebo rate (24.08%); controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 2: Comparison: Main Study: M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p = 1.000, rejective multiple test procedure — [p-value comment as in outcome 6, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 3: Comparison: Main Study: M-SD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p = 1.000, rejective multiple test procedure — [p-value comment as in outcome 6, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 4: Comparison: Integrated Study (Main + Japan Sub-Study): M-SD + M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p = 0.344, rejective multiple test procedure — [p-value comment as in outcome 6, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 5: Comparison: Integrated Study (Main + Japan Sub-Study): M-HD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p = 0.559, rejective multiple test procedure — [p-value comment as in outcome 6, analysis 1]; controlling familywise Type I error of 5% in a strong sense
Statistical Analysis 6: Comparison: Integrated Study (Main + Japan Sub-Study): M-SD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — one-sample two-sided Chi-square test; p = 0.815, rejective multiple test procedure — [p-value comment as in outcome 6, analysis 1]; controlling familywise Type I error of 5% in a strong sense

ADVERSE EVENTS:
Time Frame: See time frame specifics detailed for each reporting group in their respective descriptions below.
Description: Treatment-emergent adverse events (TEAEs) are presented.
Groups:
- Integrated Study (Main + Japan Sub- Study): I-SD: Participants randomized to receive adalimumab 2.4 mg/kg (maximum dose of 160 mg) at Baseline and matching placebo at Week 1, 1.2 mg/kg (maximum dose of 80 mg) at Week 2, followed by 0.6 mg/kg (maximum dose of 40 mg) at Week 4 and Week 6.
  TEAEs during induction period: events with an onset date on or after first dose date of study drug in induction period and up to 70 days after last dose date of the study drug in induction period and prior to first dose date of study drug in maintenance period. Mean duration of treatment was 52.8 days.
- Integrated Study (Main + Japan Sub- Study): I-HD: Participants randomized to receive adalimumab 2.4 mg/kg (maximum dose of 160 mg) at Baseline and at Week 1, 1.2 mg/kg (maximum dose of 80 mg) at Week 2, followed by 0.6 mg/kg (maximum dose of 40 mg) at Week 4 and Week 6.
  TEAEs during induction period: events with an onset date on or after first dose date of study drug in induction period and up to 70 days after last dose date of the study drug in induction period and prior to first dose date of study drug in maintenance period. Mean duration of treatment was 55.4 days.
- Integrated Study (Main + Japan Sub- Study): I-HD-OL: (After Amendment 4) participants assigned to open-label adalimumab 2.4 mg/kg (maximum dose of 160 mg) at Baseline and at Week 1, 1.2 mg/kg (maximum dose of 80 mg) at Week 2, followed by 0.6 mg/kg (maximum dose of 40 mg) at Week 4 and Week 6.
  TEAEs during induction period: events with an onset date on or after first dose date of study drug in induction period and up to 70 days after last dose date of the study drug in induction period and prior to first dose date of study drug in maintenance period. Mean duration of treatment was 53.8 days.
- Integrated Study (Main + Japan Sub- Study): M-SD: Participants demonstrating a clinical response per PMS (defined as a decrease in PMS ≥ 2 points and ≥ 30% from Baseline) at Week 8 randomized to adalimumab maintenance standard dose (0.6 mg/kg [maximum dose of 40 mg] eow). Participants were to continue their blinded treatment during the maintenance period until Week 52 unless they had ≥ 2 flares and got open label adalimumab rescue therapy after the second flare.
  TEAEs during maintenance period: events with an onset date on or after first dose date of study drug in maintenance period and prior to re-randomization due to first disease flare if applicable and up to 70 days after the last dose date of the study drug in maintenance period. Events with an onset date on or after the first dose date in long-term follow-up study M10-870 (NCT02632175) are excluded. Mean duration of treatment was 226.8 days.
- Integrated Study (Main + Japan Sub- Study): M-HD: Participants demonstrating a clinical response per PMS (defined as a decrease in PMS ≥ 2 points and ≥ 30% from Baseline) at Week 8 randomized to adalimumab maintenance high dose (0.6 mg/kg [maximum dose of 40 mg] ew). Participants were to continue their blinded treatment during the maintenance period until Week 52 unless they had ≥ 2 flares and got open label adalimumab rescue therapy after the second flare.
  TEAEs during maintenance period: events with an onset date on or after first dose date of study drug in maintenance period and prior to re-randomization due to first disease flare if applicable and up to 70 days after the last dose date of the study drug in maintenance period. Events with an onset date on or after the first dose date in long-term follow-up study M10-870 (NCT02632175) are excluded. Mean duration of treatment was 241.0 days.
- Integrated Study (Main + Japan Sub- Study): M-PL: (Prior to Amendment 4) participants demonstrating a clinical response per PMS (defined as a decrease in PMS ≥ 2 points and ≥ 30% from Baseline) at Week 8 randomized to maintenance placebo. Participants were to continue their blinded treatment during the maintenance period until Week 52 unless they had ≥ 2 flares and got open label adalimumab rescue therapy after the second flare.
  TEAEs during maintenance period: events with an onset date on or after first dose date of study drug in maintenance period and prior to re-randomization due to first disease flare if applicable and up to 70 days after the last dose date of the study drug in maintenance period. Events with an onset date on or after the first dose date in long-term follow-up study M10-870 (NCT02632175) are excluded. Mean duration of treatment was 184.2 days.
- Integrated Study (Main + Japan Sub- Study): Any Adalimumab: Participants receiving any adalimumab during Induction or Maintenance Phase.
  Any Adalimumab TEAEs: events with an onset date on or after first dose date of adalimumab and up to 70 days after the last dose date of adalimumab and prior to the first dose date in M10-870 if applicable, whichever comes first. For participants who received placebo during the maintenance period, TEAE collection period ends 70 days after last induction dose of adalimumab and re-starts with their next adalimumab dose, if applicable. Mean duration of treatment was 256.3 days.
Arm/Group | Integrated Study (Main + Japan Sub- Study): I-SD | Integrated Study (Main + Japan Sub- Study): I-HD | Integrated Study (Main + Japan Sub- Study): I-HD-OL | Integrated Study (Main + Japan Sub- Study): M-SD | Integrated Study (Main + Japan Sub- Study): M-HD | Integrated Study (Main + Japan Sub- Study): M-PL | Integrated Study (Main + Japan Sub- Study): Any Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/51 | 0/18 | 0/33 | 0/36 | 0/12 | 0/101
Serious Adverse Events (participants affected / at risk) | 5/32 | 4/51 | 1/18 | 5/33 | 5/36 | 1/12 | 22/101
Other Adverse Events (participants affected / at risk) | 13/32 | 16/51 | 14/18 | 15/33 | 20/36 | 10/12 | 65/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Integrated Study (Main + Japan Sub- Study): I-SD (N=32) | Integrated Study (Main + Japan Sub- Study): I-HD (N=51) | Integrated Study (Main + Japan Sub- Study): I-HD-OL (N=18) | Integrated Study (Main + Japan Sub- Study): M-SD (N=33) | Integrated Study (Main + Japan Sub- Study): M-HD (N=36) | Integrated Study (Main + Japan Sub- Study): M-PL (N=12) | Integrated Study (Main + Japan Sub- Study): Any Adalimumab (N=101)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (4)
PERICARDITIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 10 (11)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ENTERITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENTERITIS INFECTIOUS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
MENINGITIS ASEPTIC (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Integrated Study (Main + Japan Sub- Study): I-SD (N=32) | Integrated Study (Main + Japan Sub- Study): I-HD (N=51) | Integrated Study (Main + Japan Sub- Study): I-HD-OL (N=18) | Integrated Study (Main + Japan Sub- Study): M-SD (N=33) | Integrated Study (Main + Japan Sub- Study): M-HD (N=36) | Integrated Study (Main + Japan Sub- Study): M-PL (N=12) | Integrated Study (Main + Japan Sub- Study): Any Adalimumab (N=101)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 9 (9)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NONINFECTIVE CONJUNCTIVITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (3) | 1 (1) | 1 (1) | 6 (11)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (5)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 2 (2) | 11 (14)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
FATIGUE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PERIPHERAL SWELLING (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
PYREXIA (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
NASOPHARYNGITIS (Infections and infestations) | 2 (2) | 2 (2) | 1 (2) | 3 (4) | 4 (4) | 1 (1) | 12 (18)
PHARYNGITIS (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (3) | 9 (10)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
STREPTOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 3 (4) | 0 (0) | 2 (3) | 4 (4) | 2 (2) | 10 (13)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
JOINT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 5 (5)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MONOCYTE COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 4 (4) | 5 (7) | 4 (6) | 6 (6) | 2 (2) | 2 (2) | 19 (28)
TREMOR (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
GLYCOSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (6)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 7 (8)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
HANGNAIL (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/57/NCT02065557/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT02065557/SAP_001.pdf